CLINICAL TRIAL: NCT03315338
Title: A Phase I Adaptive Dose, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacological Effects of Orally Administered CORT118335 in Healthy Subjects
Brief Title: First-in-human Study in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CORT118335-850
Record Dates: First submitted 2017-09-27; First posted 2017-10-20 (Actual); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Healthy
MeSH Terms: interventions — CORT118335; Prednisone; Glucose

STUDY DESIGN:
Intervention Model Description: The 5 study parts may not be conducted entirely sequentially provided that this is justified by PK and safety data obtained from completed cohorts. The first MAD cohort will not start until data are available from at least 2 SAD levels using the same formulation.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (31):
- SAD Part 1 Active Cohort A (Experimental): CORT118335, 25 mg
  Interventions: Drug: CORT118335, 25 mg
- SAD Part 1 Placebo oral capsule Cohort A (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- SAD Part 1 Active Cohort B (Experimental): CORT118335, 75mg
  Interventions: Drug: CORT118335, 75mg
- SAD Part 1 Placebo Cohort B (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- SAD Part 1 Active Cohort C (Experimental): CORT118335, 225mg
  Interventions: Drug: CORT118335, 225mg
- SAD Part 1 Placebo Cohort C (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- SAD Part 1 Active Cohort D (Experimental): CORT118335, 675mg
  Interventions: Drug: CORT118335, 675mg
- SAD Part 1 Placebo Cohort D (Placebo Comparator)
  Interventions: Drug: Placebo oral capsule
- SAD Part 2 Active Cohort A, Fasting (Experimental): CORT118335, 600mg, is supplied as capsules for oral dosing given after an overnight fast
  Interventions: Drug: CORT118335, 600mg
- SAD Part 2 Active Cohort A, Fed (Experimental): CORT118335, 600mg, is supplied as capsules for oral dosing given after a high-fat breakfast
  Interventions: Drug: CORT118335, 600mg
- SAD Part 2 Placebo PD Effect Cohort B (Placebo Comparator)
  Interventions: Drug: Prednisone Oral Tablet; Drug: Glucose; Drug: Placebo oral capsule
- SAD Part 2 Active PD Effect Cohort B: 630mg of CORT118335 (Experimental)
  Interventions: Drug: Prednisone Oral Tablet; Drug: Glucose; Drug: CORT118335, 630mg
- SAD Part 2 Active PD Effect Cohort B: 675mg of CORT118335 (Experimental)
  Interventions: Drug: Prednisone Oral Tablet; Drug: Glucose; Drug: CORT118335, 675mg
- MAD Part 3 Active Cohort A (Experimental): CORT118335, 375mg qd for 14 days
  Interventions: Drug: CORT118335, 375mg
- MAD Part 3 Placebo Cohort A (Placebo Comparator): Placebo qd for 14 days
  Interventions: Drug: Placebo oral capsule
- SAD Part 4 Active Cohort A (Experimental): CORT118335, 100mg
  Interventions: Drug: CORT118335, 100mg
- SAD Part 4 Placebo Cohort A (Placebo Comparator)
  Interventions: Drug: Placebo oral suspension
- SAD Part 4 Active Cohort B (Experimental): CORT118335, 300mg
  Interventions: Drug: CORT118335, 300mg
- SAD Part 4 Placebo Cohort B (Placebo Comparator)
  Interventions: Drug: Placebo oral suspension
- SAD Part 4 Active Cohort C, Fasting (Experimental): CORT118335, 900mg is supplied as suspension for oral dosing given after an overnight fast
  Interventions: Drug: CORT118335, 900mg
- SAD Part 4 Active Cohort C, Fed (Experimental): CORT118335, 900mg is supplied as suspension for oral dosing given after a high-fat breakfast
  Interventions: Drug: CORT118335, 900mg
- SAD Part 4 Placebo Cohort C, Fasting (Placebo Comparator): Supplied as suspension for oral dosing given after an overnight fast
  Interventions: Drug: Placebo oral suspension
- SAD Part 4 Placebo Cohort C, Fed (Placebo Comparator): Supplied as suspension for oral dosing given after a high-fat breakfast
  Interventions: Drug: Placebo oral suspension
- SAD Part 4 Active Cohort Part D (Experimental): CORT118335, 1500mg
  Interventions: Drug: CORT118335, 1500mg
- SAD Part 4 Placebo Cohort D (Placebo Comparator)
  Interventions: Drug: Placebo oral suspension
- MAD Part 5 Active Cohort A (Experimental): CORT118335, 150mg
  Interventions: Drug: CORT118335, 150mg
- MAD Part 5 Placebo Cohort A (Placebo Comparator)
  Interventions: Drug: Placebo oral suspension
- MAD Part 5 Active Cohort B (Experimental): CORT118335, dose to be determined
  Interventions: Drug: CORT118335, dose to be determined
- MAD Part 5 Placebo Cohort B (Placebo Comparator)
  Interventions: Drug: Placebo oral suspension
- MAD Part 5 Active Cohort C (Experimental): CORT118335, dose to be determined
  Interventions: Drug: CORT118335, dose to be determined
- MAD Part 5 Placebo Cohort C (Placebo Comparator)
  Interventions: Drug: Placebo oral suspension

INTERVENTIONS:
Drug: CORT118335, 25 mg — CORT118335 is supplied as capsules for oral dosing
  Arms: SAD Part 1 Active Cohort A
Drug: Prednisone Oral Tablet — Challenge Agent, Dose and Route of Administration:
  Standard release 1x20mg and 1x5mg (25mg total) dose, orally administered.
  Arms: SAD Part 2 Active PD Effect Cohort B: 630mg of CORT118335; SAD Part 2 Active PD Effect Cohort B: 675mg of CORT118335; SAD Part 2 Placebo PD Effect Cohort B
Drug: Glucose — 75 g in 300 mL solution, orally administered
  Arms: SAD Part 2 Active PD Effect Cohort B: 630mg of CORT118335; SAD Part 2 Active PD Effect Cohort B: 675mg of CORT118335; SAD Part 2 Placebo PD Effect Cohort B
Drug: Placebo oral suspension — Reference Therapy, Dose and Route of Administration:
  Placebo suspension, orally administered.
  Arms: MAD Part 5 Placebo Cohort A; MAD Part 5 Placebo Cohort B; MAD Part 5 Placebo Cohort C; SAD Part 4 Placebo Cohort A; SAD Part 4 Placebo Cohort B; SAD Part 4 Placebo Cohort C, Fasting; SAD Part 4 Placebo Cohort C, Fed; SAD Part 4 Placebo Cohort D
Drug: CORT118335, 75mg — CORT118335 is supplied as capsules for oral dosing
  Arms: SAD Part 1 Active Cohort B
Drug: CORT118335, 225mg — CORT118335 is supplied as capsules for oral dosing
  Arms: SAD Part 1 Active Cohort C
Drug: CORT118335, 675mg — CORT118335 is supplied as capsules for oral dosing
  Arms: SAD Part 1 Active Cohort D; SAD Part 2 Active PD Effect Cohort B: 675mg of CORT118335
Drug: CORT118335, 600mg — CORT118335 is supplied as capsules for oral dosing
  Arms: SAD Part 2 Active Cohort A, Fasting; SAD Part 2 Active Cohort A, Fed
Drug: CORT118335, 630mg — CORT118335 is supplied as capsules for oral dosing
  Arms: SAD Part 2 Active PD Effect Cohort B: 630mg of CORT118335
Drug: CORT118335, 375mg — CORT118335 is supplied as capsules for oral dosing
  Arms: MAD Part 3 Active Cohort A
Drug: CORT118335, 100mg — CORT118335 is supplied as a suspension for oral dosing
  Arms: SAD Part 4 Active Cohort A
Drug: CORT118335, 300mg — CORT118335 is supplied as a suspension for oral dosing
  Arms: SAD Part 4 Active Cohort B
Drug: CORT118335, 900mg — CORT118335 is supplied as a suspension for oral dosing
  Arms: SAD Part 4 Active Cohort C, Fasting; SAD Part 4 Active Cohort C, Fed
Drug: CORT118335, 150mg — CORT118335 is supplied as a suspension for oral dosing
  Arms: MAD Part 5 Active Cohort A
Drug: CORT118335, 1500mg — CORT118335 is supplied as a suspension for oral dosing
  Arms: SAD Part 4 Active Cohort Part D
Drug: Placebo oral capsule — Placebo capsules, orally administered
  Arms: MAD Part 3 Placebo Cohort A; SAD Part 1 Placebo Cohort B; SAD Part 1 Placebo Cohort C; SAD Part 1 Placebo Cohort D; SAD Part 1 Placebo oral capsule Cohort A; SAD Part 2 Placebo PD Effect Cohort B
Drug: CORT118335, dose to be determined — CORT118335 is supplied as suspension for oral dosing
  Arms: MAD Part 5 Active Cohort B; MAD Part 5 Active Cohort C

SUMMARY:
This initial Phase I study will evaluate the safety, tolerability, and pharmacokinetics (PK) of single and multiple ascending doses of CORT118335, the effect of concomitant administration with food on exposure to CORT118335, and its pharmacological effect in healthy subjects.

DETAILED DESCRIPTION:
This is a 5-part, single-center study of single and multiple ascending doses of CORT118335 in healthy subjects.

Parts I and 4 of the study are double-blind, randomized, placebo-controlled assessments of single-ascending doses (SAD) of CORT118335. Subjects will be enrolled sequentially into 1 of up 8 cohorts (Part 1, Cohorts A to D [Cohorts E to G have been cancelled]; Part 4, Cohorts A to D), each containing 8 subjects. Within each cohort, 6 subjects will be randomly assigned to receive a single dose of CORT118335 and 2 subjects will be randomly assigned to receive a single dose of matching placebo.

Part 2 Cohort A, food-effect, will be an open-label 2-way crossover study in one cohort of 12 subjects, randomized in a 1:1 ratio to receive a single dose of CORT118335 once after an overnight fast and once after a high-fat breakfast or the alternate sequence, over 2 study periods separated by a washout of at least 7 days/5 half-lives.

Part 2 Cohort B, PD cohort, will be a double-blind, randomized, placebo-controlled, 3-way cross-over study and will serve as proof of pharmacological effect (GR modulation) for CORT118335. Subjects will be randomized in a 1:1:1 ratio to receive placebo, and two dose levels of CORT118335 in one of three treatment sequences across 3 study periods separated by washouts of at least 7 days/5 half-lives. On each occasion, the ability of CORT118335 to ameliorate the pharmacological effects of a single dose of prednisone will be measured.

Parts 3 and 5 are double-blind, randomized, placebo-controlled assessments of multiple oral ascending doses of CORT118335. Subjects will be enrolled sequentially into 1 of up to 4 cohorts (Part 1 Cohort A [Cohorts B to D have been cancelled; Part 5 Cohorts A to C), each containing 12 subjects. Within each cohort, 9 subjects will be randomly assigned to receive CORT118335 and 3 subjects to receive matching placebo daily for 14 days.

Different formulations of CORT118335 will be used in Parts 1, 2 and 3, and in Parts 4 and 5.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects or non-pregnant, non-lactating healthy female subjects of non-childbearing potential
* Age 18 to 60 years
* Body mass index (BMI) of 18.0 to 30.0 kg/m2
* Weight of ≤102 kg
* Must be willing and able to communicate and participate in the whole study
* Morning serum cortisol of 5 μg/dL to 23 μg/dL (138 nmol/L to 635 nmol/L) at screening and/or Day -1 for multiple dose cohorts
* Must provide written informed consent
* Must agree to use an adequate method of contraception
* Must agree to adhere to study restrictions

Exclusion Criteria:

* Subjects who have received any IMP in a clinical research study within the 3 months before the first dose in this study
* Subjects who are study site or Sponsor employees, or immediate family members of a study site or Sponsor employee
* Subjects who have previously been enrolled in this study
* Males who have a pregnant partner
* History of any drug or alcohol abuse in the year before the first dose in this study
* Regular alcohol consumption in male subjects >21 units per week and female subjects >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Current smokers and those who have smoked within the 6 months before the first dose in this study. A breath carbon monoxide reading of greater than 10 ppm at screening or on admission
* Current users of e-cigarettes and nicotine replacement products and those who have used these products within the 6 months before the first dose in this study
* Subjects who do not have suitable veins for multiple venepunctures/cannulation as assessed by the Investigator at screening
* Clinically significant abnormal biochemistry, hematology or urinalysis as judged by the Investigator
* Positive drugs of abuse test result at screening or on admission (amphetamines, barbiturates, benzodiazepines, cocaine, marijuana/cannabis, methadone, methamphetamine/ecstasy, morphine/opiates, phencyclidine, tricyclic antidepressants)
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* Subject has active renal and/or hepatic disease, as evidenced by:

  * an estimated glomerular filtration rate (eGFR) of <60 mL/min/1.73m2 using Modification of Diet in Renal Disease (MDRD) equation at screening
  * ALT and/or AST >1.5 times the upper limit of normal at screening or on admission
  * subjects with borderline results can have these tests repeated once.
* History of clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, respiratory, gastrointestinal or neurological disease as judged by the Investigator
* Subject had any form of cancer within the 2 years before first dose in this study*, with the exception of basal cell and/or squamous cell cancer of the skin that has been treated completely and is without evidence of local recurrence or metastasis
* Subject has a history and/or symptoms of adrenal insufficiency
* Subject has consumed liquorice or other glycyrrhetic acid derivatives regularly, in the judgement of the Investigator, in the 6 months before the first dose of study medication
* Subject has a history of jaundice and/or subject has had a cholecystectomy
* Subject has a history of clinically significant gastrointestinal disease including gastroesophageal reflux disease, malabsorption syndrome, colon cancer, chronic colitis, Crohn's disease, inflammatory bowel disease, gastroparesis, constipation, chronic diarrhoea, obstruction, gastrointestinal bleeding, and/or peptic ulcers
* Subject has a condition that could be aggravated by glucocorticoid and/or mineralocorticoid blockade (e.g., asthma, any chronic inflammatory condition) or activation (e.g., immunodeficiency, active infection)
* Subjects with inactive seasonal hay fever may be included. Subjects with childhood (aged less than 18 years) asthma may be included provided they have had no symptoms and required no treatment for at least 5 years
* Subjects with a QTcF interval of >450 msec at screening or pre-dose, based on the mean of three ECGs
* History of additional risk factors for torsades de pointes (e.g., heart failure, hypokalaemia, family history of long QT syndrome)
* Supine heart rate at rest of <40 bpm or >100 bpm. BP out with the following ranges: diastolic BP 40-90; systolic BP 90-140 (subjects aged 18-45 year) and 90-160 (subjects aged >45 year). Heart rate and blood pressure can be retested twice in the supine position at intervals of 5 min on a given day at screening and admission.
* Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients including glucose/fructose intolerance for the standard oral glucose tolerance test (OGTT)
* Presence or history of clinically significant allergy requiring treatment, as judged by the Investigator.
* Donation or loss of greater than 400 mL of blood within the 3 months before first study dose
* Subjects who are taking, or have taken, any prescribed, over-the-counter drug (other than 4 g per day paracetamol) or herbal remedies within 14 days, or for which 5 times the medication's elimination half-life will not be completed if longer, before the first dose of study medication. Exceptions may apply on a case by case basis, if considered not to interfere with the objectives of the study, as agreed by the Investigator and Sponsor's medical monitor. Standard dose multivitamins are permitted throughout the study period
* Subjects who are currently using glucocorticoids or have a history of systemic glucocorticoid use at any dose within the last 12 months or 3 months for inhaled products
* Subjects who are taking, or have taken enzyme inducers within 30 days before the first dose of study medication
* Subject is expected to require use of any medication (with the exception of standard dose multivitamins) during the study period
* Subject has a history or presence of any medical condition or disease which, in the opinion of the Investigator, could interfere with the conduct of the study or could put the subject at unacceptable risk. This specifically includes any subject with flu or flu-like symptoms
* Failure to satisfy the Investigator of fitness to participate for any other reason

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 143 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-02-22 (Actual); Study Completion 2019-02-22 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | SAD Cohorts: Day -28 to Day 7; Part 2A Cohorts: Day -28 to Day 14; Part 2B Cohorts: Day -28 to Day 21; MAD Cohorts: Day -28 to Day 21

SECONDARY OUTCOMES:
QT interval corrected for heart rate using Fridericia's formula (QTcF) exposure-response analysis | SAD parts: Pre dose through 24 hours post dose. MAD parts: Pre first dose through 24 hours post final dose of Investigational Medicinal Product (IMP
tlag Pharmacokinetic (PK) parameter | SAD parts: Pre dose through 96 hours post dose; MAD parts: Pre first dose through 96 hours post final dose of IMP
  The elapsed time from dosing at which analyte was first quantifiable in a concentration vs time profile (tlag)
tmax PK parameter | SAD parts: Pre dose through 96 hours post dose; MAD parts: Pre first dose through 96 hours post final dose of IMP
  The time from dosing at which Cmax was apparent (tmax)
Cmax PK parameter | SAD parts: Pre dose through 96 hours post dose; MAD parts: Pre first dose through 96 hours post final dose of IMP
  Maximum observed concentration (Cmax)
tmin (MAD only) PK parameter | MAD parts: Pre first dose through 96 hours post final dose of IMP
  Time from dosing of the minimum plasma drug concentration (tmin)
Cmin (MAD only) PK parameter | MAD parts: Pre first dose through 96 hours post final dose of IMP
  Minimum plasma drug concentration (Cmin)
Clast PK parameter | SAD parts: Pre dose through 96 hours post dose; MAD parts: Pre first dose through 96 hours post final dose of IMP
  Last measurable concentration (Clast)
tlast PK parameter | SAD parts: Pre dose through 96 hours post dose; MAD parts: Pre first dose through 96 hours post final dose of IMP
  Time from dosing of the last measurable concentration (tlast)
t1/2 PK parameter | SAD parts: Pre dose through 96 hours post dose; MAD parts: Pre first dose through 96 hours post final dose of IMP
  The apparent elimination half-life (t1/2)
lambda-z PK parameter | SAD parts: Pre dose through 96 hours post dose; MAD parts: Pre first dose through 96 hours post final dose of IMP
  The slope of the apparent elimination phase (lambda-z)
AUCinf PK parameter | SAD parts: Pre dose through 96h post dose; MAD parts: Pre first dose through 96h post final dose of IMP
  Area under the plasma concentration-time curve from time zero to infinity (AUCinf)
AUC(0-last) PK parameter | SAD parts: Pre dose through 96 hours post dose; MAD parts: Pre first dose through 96 hours post final dose of IMP
  Area under the curve from 0 time to last measurable concentration [AUC(0-last)]
AUC(0-24) PK parameter | SAD parts: Pre dose through 24 hours post dose; MAD parts: Pre first dose through 24 hours post final dose of IMP
  Area under the curve from 0 time to 24 h post dose [AUC(0-24)]
Food effect: AUC(0-last) PK parameter | Pre first dose through 96 hours post final dose
Food effect: AUC(0-inf) PK parameter | Pre first dose through 96 hours post final dose
  Area under the curve from 0 time extrapolated to infinity [AUC(0-inf)]
Food effect: Cmax PK parameter | Pre first dose through 96 hours post final dose
Pharmacodynamics (PD): peripheral differential white blood cell count | Pre first dose through 24 hours post final dose
PD: serum osteocalcin and adiponectin concentrations | Pre first dose through 24 hours post final dose
PD: messenger ribonucleic acid (mRNA) expression for selected genes in whole blood | Pre first dose through 24 hours post final dose
PD: glucose tolerance | Pre first dose through 24 hours post final dose
Homeostatic model assessment of insulin-resistance (HOMA-IR) | Pre-dose through Day 14

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Mair, MBChB, MFPM, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided